CLINICAL TRIAL: NCT05861674
Title: A Multicenter, Randomized, Controlled, Open-label Phase IIb Study to Assess Efficacy and Safety of HH-003 Injection in Subjects With Chronic Hepatitis Delta Virus Infection
Brief Title: A Study to Assess Efficacy and Safety of HH-003 Injection in Subjects With Chronic Hepatitis Delta Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH003-204
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis Delta Virus Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HH-003 (20mg/kg)+TAF (Experimental): Subjects will receive HH-003 20 mg/kg Q2W intravenously and TAF 25 mg QD orally during 48-week treatment period, and receive TAF 25 mg QD orally during 24-week follow-up period.
  Interventions: Biological: HH-003(20mg/kg); Drug: TAF
- HH-003 (10mg/kg)+TAF (Experimental): Subjects will receive HH-003 10 mg/kg Q2W intravenously and TAF 25 mg QD orally during 48-week treatment period, and receive TAF 25 mg QD orally during 24-week follow-up period.
  Interventions: Biological: HH-003(10mg/kg); Drug: TAF
- TAF (Other): Subjects will receive TAF 25 mg QD orally during 48-week treatment period and 24-week follow-up period.
  Interventions: Drug: TAF

INTERVENTIONS:
Biological: HH-003(20mg/kg) — 20 mg/kg Q2W intravenously for 48 weeks
  Arms: HH-003 (20mg/kg)+TAF
Biological: HH-003(10mg/kg) — 10 mg/kg Q2W intravenously for 48 weeks
  Arms: HH-003 (10mg/kg)+TAF
Drug: TAF — TAF 25 mg QD orally during 48-week treatment period and 24-week follow-up period

SUMMARY:
This is a multicenter, randomized, controlled, open-label, Phase IIb study of HH-003 injection, HH-003 injection is a monoclonal antibody targeting Hepatitis B virus. This study aims to assess efficacy and safety in subjects with chronic hepatitis delta virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form;
* Male or female aged 18 to 70 years;
* Positive HBsAg at screening;
* History of chronic HDV infection for at least 6 months prior to randomization. For subjects also recommended for anti-HBV therapy, previous first line NrtIs treatment (ETV, TDF, TAF) within at least 12 weeks prior to the planned start of study treatment or subject's willingness to take first line NrtIs treatment for at least 12 weeks prior to the planned start of study treatment is required;
* Positive HDV antibody at screening;
* HDV RNA ≥100 IU/mL at screening;
* 1×ULN<Alanine aminotransferase (ALT) <10×ULN at screening;

Exclusion Criteria:

* Subjects with known hypersensitivity to HH-003 and its components, history of severe allergic reaction to other therapeutic antibodies or severe allergic diseases;
* Subjects with contraindications for TAF;
* History of interferon therapy within 3 months before randomization;
* Any of the following lab test results at screening:

  1. Total bilirubin >2×ULN (except for subjects with Gilbert syndrome);
  2. Direct bilirubin > 1.5×ULN ;
  3. Platelets<80,000/mm3 (80×109/L);
  4. Serum Albumin <35 g/L;
  5. Prothrombin time international normalized ratio (INR) >1.3;
  6. Hemoglobin <100 g/L;
  7. Absolute neutrophils<1,500/mm3 (1.5×109/L);
  8. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 (according to the calculation equation of CKD-MDRD);
* Concomitant decompensated cirrhosis (cirrhosis with complications of portal hypertension and/or decreased hepatic function). The diagnosis of cirrhosis is based on, but not limited to: liver imaging assessment within 6 months prior to randomization (including screening period) (e.g.: liver ultrasound) or cirrhosis indicated by histopathology of liver biopsy, or liver stiffness measurement LSM≥17 kPa at screening, refer to more serious reported findings;
* Hepatic insufficiency within 3 months prior to randomization (including but not limited to: ascites, hepatic encephalopathy, upper gastrointestinal hemorrhage);
* Previous or current hepatocellular carcinoma (HCC) or suspicion for HCC suggested by liver histopathology or liver imaging; or serum alpha-fetoprotein (AFP) ≥ 50 ng/mL at screening;
* Subjects with history of alcoholic liver disease, nonalcoholic steatohepatitis, autoimmune liver disease or other hereditary liver diseases, drug-induced liver disease or other clinically significant chronic liver diseases not caused by HDV/HBV;
* History of other malignancies other than HCC, unless the subject's malignancy has been in complete remission within 3 years prior to screening and does not require chemotherapy and additional medical or surgical intervention; invasive medical devices within 1 month before randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with serum HDV RNA below the lower limit of detection or a decrease of ≥2 log10 IU/mL from baseline and ALT normalization | At Week 24 of the treatment period

SECONDARY OUTCOMES:
Proportion of subjects with serum HDV RNA below the lower limit of detection or a decrease of ≥2 log10 IU/mL from baseline | At Week 24 of the treatment period
Proportion of subjects with ALT normalization | At Week 24 of the treatment period
Change from baseline in liver stiffness measurement (LSM) | At Week 24 of the treatment period
Proportion of subjects with serum HDV RNA below the lower limit of detection or a decrease of ≥2 log10 IU/mL from baseline and ALT normalization | At Week 48 of the treatment period
Proportion of subjects with serum HDV RNA below the lower limit of detection or a decrease of ≥2 log10 IU/mL from baseline | At Week 48 of the treatment period
Proportion of subjects with ALT normalization | At Week 48 of the treatment period
Change from baseline in liver stiffness measurement (LSM) | At Week 48 of the treatment period
Proportion of subjects with serum HDV RNA below the lower limit of detection or a decrease of ≥2 log10 IU/mL from baseline | At Week 24 of the follow-up period
Proportion of subjects with ALT normalization | At Week 24 of the follow-up period
Change from baseline in liver stiffness measurement (LSM) | At Week 24 of the follow-up period
Change from baseline in serum HDV RNA levels at different time points | Up to Week 72
Change from baseline in serum ALT levels at different time points | Up to Week 72

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital Captial Medical University, Beijing, Beijing Municipality, China